CLINICAL TRIAL: NCT04349969
Title: A Phase 1 Multicenter, Open Label, Dose Escalation and Dose Expansion Study to Evaluate the Safety, Pharmacokinetics, and Antitumor Activity of AK117 as Monotherapy or in Combination With AK104 in Subjects With Relapsed/Refractory Advanced or Metastatic Solid Tumors or Lymphomas
Brief Title: A Study to Evaluate the Safety, Pharmacokinetics, and Antitumor Activity of AK117 as Monotherapy or in Combination With AK104
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Akesobio Australia Pty Ltd (Industry)
Responsible Party: Sponsor
Organization: Akeso (Industry)
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: AK117-101
Record Dates: First submitted 2020-04-14; First posted 2020-04-16 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Neoplasms Malignant
Keywords: Antineoplastic Agents, Immunological
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): Parts A and B: AK117 monotherapy intravenous (IV) infusion- weekly doses in a 28-day cycle.
  Parts A2: AK117 (QW) + AK104 (Q3W) combination therapy intravenous (IV) infusion in a 21-day cycle.
  Interventions: Drug: AK117; Drug: AK117+AK104

INTERVENTIONS:
Drug: AK117 — All subjects will receive 4 weekly infusions (Days 1, 8, 15, and 22) of AK117 in each 28-day treatment cycle until unacceptable toxicity, documentation of confirmed progressive disease (PD), or subject withdrawal.
Drug: AK117+AK104 — All Subjects will receive 3 weekly infusions of AK117 (Days 1, 8, and 15) and 1 infusion of AK104 (on Day 1) as combination therapy in each 21-day treatment cycle until unacceptable toxicity, documentation of confirmed PD, or subject withdrawal.

SUMMARY:
This was a first-in-human, Phase 1 study designed to evaluate the safety, tolerability, PK, immunogenicity, pharmacodynamics, and preliminary antitumor activity of AK117 as monotherapy or in combination with AK104 in subjects with advanced or metastatic solid tumors.

DETAILED DESCRIPTION:
The study was conducted across 2 parts. Part A of the study was the dose escalation part of AK117 monotherapy as priming dose to evaluate the safety and tolerability of AK117 weekly dosing in solid tumors. Part B which was to evaluate the optimal maintenance dose of AK117 was not performed as the MAD dose level of AK117 monotherapy was determined in Part A.

Part A2 was the dose escalation part of AK117 in combination with AK104 to evaluate the safety and tolerability of AK117 monotherapy in solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Able to provide written and signed informed consent
2. Eastern Cooperative Oncology Group (ECOG) performance status (PS) score of 0 or 1.
3. Life expectancy ≥12 weeks
4. Females of childbearing potential and non-sterilized males who are sexually active must use an effective method of contraception from screening until 120 days after final dose of investigational product or women of non-childbearing potential.
5. Willing to receive blood transfusion(s) when so advised by the investigator.
6. Adequate organ function.
7. Subjects must have a histologically or cytologically confirmed advanced solid tumor that is refractory or relapsed to the current standard therapies or which no effective standard therapy is available.
8. At least 1 measurable lesion according to RECIST v1.1

Exclusion Criteria:

1. Concurrent enrollment in another clinical study excluding observational trials
2. Prior malignancy active within the previous 3 years except for the tumor for which a subject is enrolled in the study
3. Active brain/central nervous system (CNS) metastases
4. Active infections requiring systemic therapy within 2 weeks prior to the first dose of investigational product.
5. Known history of HIV.
6. Known active hepatitis B or C infections
7. Active or prior documented autoimmune disease that may relapse.
8. History of interstitial lung disease or non-infectious pneumonitis, except those induced by radiation therapies.
9. History of defects in RBC production, or hemoglobin production or metabolism
10. Patients with clinically significant cardio-cerebrovascular disease.
11. History of severe hypersensitivity reactions to other mAbs.
12. History of organ transplantation.
13. Receiving any anticancer therapy targeting the CD47/SIRPα ; Anticancer small molecule targeted agent within 2 weeks prior to the first dose of the investigational product; Anticancer mAbs within 6 weeks prior to the first dose of investigational product or 5 half-lives (whichever is lesser); Other anticancer therapy within 4 weeks prior to the first dose of the investigational product;
14. Subjects with a condition requiring systemic treatment with either corticosteroid (>10 mg daily doses)) or other immunosuppressive medications within 2 weeks prior to the first dose of investigational product.
15. Received a live attenuated vaccine within 4 weeks prior to the first dose of investigational product.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2020-04-23 (Actual); Primary Completion 2022-11-08 (Actual); Study Completion 2022-11-08 (Actual)

PRIMARY OUTCOMES:
Incidence and nature of adverse events (AEs) | From the time of informed consent signed through 30 days after the last dose of AK117 as monotherapy or in combination with AK104
  An AE is defined as any untoward medical occurrence in a participant administered a pharmaceutical product temporally associated with the use of study treatment, whether or not considered related to the study treatment.
Number of participants with a Dose Limiting Toxicity (DLT) | During the first 4 weeks of first treatment dose of AK117 as monotherapy or during the first 3 weeks of treatment dose of AK117+AK104 as combination therapy.
  DLTs will be assessed during the first 4 weeks (AK117 monotherapy) or first 3 weeks (AK117+AK104 combination therapy) of treatment for dose-escalation phase and are defined as toxicities that meet pre-defined severity criteria, and assessed as having a suspected relationship to study drug, and unrelated to disease, disease progression, inter-current illness, or concomitant medications that occurs within the first cycle of treatment.

SECONDARY OUTCOMES:
Objective response rate (ORR) | Up to 2 years
  ORR defined as the proportion of subjects who achieves a best overall response of CR or PR, assessed by Investigator per RECIST Version 1.1.
Disease control rate (DCR) | Up to 2 years
  (subjects achieving SD will be included in the DCR if they maintain SD for 16 and 24 weeks respectively).
Maximum observed concentration (Cmax) of AK117 as monotherapy or in combination with AK104 and Minimum observed concentration (Cmin) of AK117 at steady stateconcentration (Cmin) of AK117 at steady state | From first dose through to 30 days after last dose of investigational products.
  The endpoints for assessment of PK of AK117 and AK104 include serum concentrations of AK117 and AK104 at different timepoints after AK117 and AK104 administration.
Number of subjects who develop detectable anti-drug antibodies (ADAs) of AK117 as monotherapy or in combination with AK104 | From first dose through to 30 days after last dose of investigational products.
  The immunogenicity of AK117 and AK104 will be assessed by summarizing the number of subjects who develop detectable anti-drug antibodies (ADAs).
Area under the curve (AUC) of AK117 as monotherapy or in combination with AK104 for assessment of pharmacokinetics | From first dose through to 30 days after last dose of investigational products.
  The endpoints for assessment of PK of AK117 and AK104 include serum concentrations of AK117 and AK104 at different timepoints after AK117 and AK104 administration.
Receptor occupancy (RO) of AK117 as monotherapy or in combination with AK104 to evaluate target engagement | From first dose through to 30 days after last dose of investigational products.
  The endpoints will be measured using a flow cytometry-based method on circulating red and white blood cells.

CONTACTS AND LOCATIONS:
Locations (4):
- Australia (4):
  - Blacktown Hospital, Sydney, New South Wales
  - ICON Cancer Foundation, South Brisbane, Queensland
  - Ashford Cancer Centre Research, Kurralta Park, South Australia
  - Austin Health, Heidelberg, Victoria

IPD SHARING:
Plan to Share IPD: No